CLINICAL TRIAL: NCT01681823
Title: Phase III, Single-Center, Open Label, Trial Evaluating the Safety and Efficacy of PectaSol-C Modified Citrus Pectin on PSA Kinetics in Prostate Cancer in the Setting of Serial Increases in PSA
Brief Title: Effect of Modified Citrus Pectin on PSA Kinetics in Biochemical Relapsed PC With Serial Increases in PSA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EcoNugenics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMC12192-12CTIL
Record Dates: First submitted 2012-09-06; First posted 2012-09-10 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Prostatic Neoplasms
Keywords: Prostate Cancer; Prostatic Neoplasms; Prostate Specific Antigen; Modified Citrus Pectin; PectaSol-C; Biochemical Relapse
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Dietary Supplement: PectaSol-C Modified Citrus Pectin (MCP) Oral administration of PectaSol-C MCP (4.8 grams in six capsules three times a day away from food).
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PectaSol-C Modified Citrus Pectin (MCP) (Experimental): Treatment with 4.8 grams PectaSol-C Modified Citrus Pectin three times a day, away from meals for six months.
  Interventions: Dietary Supplement: PectaSol-C Modified Citrus Pectin (MCP)

INTERVENTIONS:
Dietary Supplement: PectaSol-C Modified Citrus Pectin (MCP) — Oral administration of PectaSol-C MCP (4.8 grams in six capsules three times a day away from food).

SUMMARY:
To determine if the oral administration of PectaSol-C Modified Citrus Pectin (MCP) is effective at improving Prostate Specific Antigen (PSA) kinetics in men with biochemical relapsed prostate cancer and serial increases in PSA levels. Also, documentation of any side effects or benefits within parameter of the study is included.

DETAILED DESCRIPTION:
This study on the effect of PectaSol-C Modified Citrus Pectin (MCP) with subjects selected on the basis of documented PC post local therapy, and biochemical relapse, with linear progression of at least 3 PSA tests in at least 3 months. After initial screening, treatment {4.8 grams (6 capsules) three times a day away from meals} will continue for 6 months provided patients are showing benefit and tolerating the therapy well. Patient tolerability of MCP will be assessed by comparing the results of monthly self-assessment diaries with baseline assessments.

Prostate cancer is the most common cancer among men, except for non melanoma skin cancer. It is the second leading cause of cancer related death in men. About 33% of prostate cancer patients treated with primary therapy (surgery or radiation) will recur in the form of non metastatic biochemically relapsed prostate cancer (BRPC-M0). In these patients, PSA is rising while scans are negative for metastasis. Recent surveys demonstrated that approximately 40% of prostate cancer patients use various complementary and alternative medicine modalities as a component of therapy. Currently, there is no standard treatment for biochemical failure with proven benefits. Patients are being encouraged to enroll in clinical trials to help establish standards of care. Studies have shown that in 80% of patients with BRPC-M0, PSA will rise by at least 25% every 6 months.

Native pectin is a complex carbohydrate soluble fiber. Dietary fibers, such as pectin, have been shown to have positive effects on a wide spectrum of pathological conditions. Their positive influence on human health is explained by their antioxidative, hypocholesterolemic, and anticancer effects. MCP is composed of short, slightly-branched, carbohydrate chains derived from the soluble albedo fraction of citrus fruit peels, which have been altered by decreasing the molecular weight and degree of esterification using pH, temperature, and a controlled enzymatic process. This specific modification is critical as it allows for the absorption of MCP into the circulatory system and ensures its targeted bioactivity throughout the body. MCP is relatively rich in galactose and thus antagonizes the binding protein galectin-3 which results in suppression of cancer cell aggregation, adhesion, and metastasis. MCP acts as a ligand for galectin-3, which plays a major role in tumor formation and progression. It has been shown using a combination of fluorescence microscopy, flow cytometry, and atomic force microscopy, that pectin galactan specifically binds to the recombinant form of human galectin-3.

MCP showed anti-metastatic effects on cancer cells in multiple in vitro and in vivo studies. MCP inhibits carbohydrate mediated tumor growth, angiogenesis and metastasis via effects on galectin-3 function as demonstrated in an animal study on MCP's inhibition of breast and colon cancer progression. Results demonstrated a 70.2% reduction in breast tumor growth, a 66% reduction in breast angiogenesis, and 0% breast to lung metastasis compared to 100% in the control group; 0% colon to liver metastasis compared to 60% in the control group; and 25% colon to lymph metastasis compared to 100% in the control group. In an earlier study oral intake of MCP had been shown to act as a potent inhibitor of spontaneous prostate carcinoma metastasis in an animal model, demonstrating a significant 56% reduction in lung metastases. Human cancer cell lines (LNCaP androgen dependent & PC3 androgen independent) and mouse prostate cancer cell lines (CASP2-1 androgen dependent and CASP1-1 androgen independent) treated with 1% MCP showed the following cytotoxicity due to induced apoptosis: 52.28% in LNCaP; 48.16% in PC3; 23.03% in CASP2-1; and 49.01% in CASP1-1.13 The effects of MCP on cell-cell and cell-matrix interactions mediated by carbohydrate-recognition were investigated by looking at MCP-inhibited B16-F1 melanoma cells adhesion and aggregation. MCP was shown to inhibit anchorage-independent growth of B16-F1 cells. These results indicate that carbohydrate-recognition by cell surface galectin-3 is involved in cell-extracellular matrix interaction and plays a role in anchorage-independent growth as well as the in vivo embolization of tumor cells. The modulation of the lung colonization of B16-F1 melanoma cells by MCP was first observed in 1992 when injection of MCP significantly decreased B16-F1 experimental metastasis (greater than 90%). Galectin-3 participation in the adhesion of the MDA-MB-435 cells to the endothelium was observed by the clustering of galectin-3 on endothelial cells at the sites of the contact with tumor cells, suggesting its potential functional significance for anti-adhesive therapy of cancer metastasis. The anti-metastatic effect of MCP has also been shown in reduced liver metastasis in a dose-dependent manner. The use of MCP in combination with the chemotherapy drug doxorubicin has demonstrated an increased cytotoxicity effect of inducing rapid cell death in prostate cancer cell lines DU-145 (androgen independent) through apoptosis, and in LNCaP (androgen dependant) through cell cycle arrest (G2-M arrest). These results show promise for the use of MCP with doxorubicin as an adjuvant to chemotherapy which may allow for lower dosage of the cancer drug to be used with less toxicity. A human clinical pilot trial with MCP showed an increase in prostate specific antigen doubling time, a marker of slowing the progression of prostate cancer. Clinical research on MCP also demonstrated a significant improvement in quality of life and stabilization of disease for patients with advanced solid tumors.

In addition to its therapeutic roles against cancer, MCP has been shown to remove toxic metals from the body without affecting essential minerals. In a clinical study, baseline levels of heavy metals and essential minerals were established with 24-hours urine collection prior to oral administration of MCP. 24-hours urine collection was repeated on days 1 and 6. Urinary excretion of lead, mercury, cadmium, and arsenic increased significantly, essential minerals were not changed significantly and no side effects were reported. In a hospital study in China, children with lead toxicity were given MCP. Their blood serum levels went down while corresponding lead levels in their urine increased significantly, without side effects.

MCP has immunostimulatory properties as demonstrated in human blood samples, including the activation of functional NK cells against K562 leukemic cells in culture: Unsaturated oligogalacturonic acids appear to be the immunostimulatory carbohydrates in MCP. Human blood samples collected from healthy volunteers were incubated with increasing concentrations of MCP and antibodies. After 24-hours, blood-antibody mix was lysed and run on a flow cytometer using a 3-color protocol and the % of activated T-cytotoxic cell subset, B-cell, and NK-cells, and % increase over untreated control calculated and a significant dose dependent activation was seen. The ability of the activated NK cells to induce leukemia cell death was analyzed by co-incubating MCP-treated lymphocytes with K562 T-cell leukemia cells and induced leukemia cell death was determined to be greater than 50%.

MCP has been demonstrated to be protective in experimental nephropathy with modulation of early proliferation and later galectin-3 expression, apoptosis and fibrosis by experimentally modulating galectin-3 in folic acid (FA)-induced acute kidney injury. Mice were pre-treated with normal or 1% MCP-supplemented drinking water one week before FA injection. During the initial injury phase, all FA treated mice lost weight whilst their kidneys enlarged secondary to the renal insult; these gross changes were significantly lessened in the MCP group but this was not associated with significant changes in galectin-3 expression. At a histological level, MCP clearly reduced renal cell proliferation but did not affect apoptosis. Later, during the recovery phase at two weeks, MCP-treated mice demonstrated reduced galectin-3 in association with decreased renal fibrosis, macrophages, proinflammatory cytokine expression and apoptosis. Galectin-3 inhibition by MCP was demonstrated to block Aldosterone (Aldo) induced collagen type I synthesis. Rats were treated with Aldo-salt combined MCP for 3 weeks. Hypertensive Aldo-treated rats presented vascular hypertrophy, inflammation, fibrosis, and increased aortic Gal-3 expression. MCP treatment reversed all the above effects.

MCP is affirmed as GRAS (generally regarded as safe) under the US Code of Federal Regulation 21CFR184.1588.

ELIGIBILITY:
Inclusion Criteria:

* Documented PC post local therapy with undetectable Prostate Specific Antigen (PSA), and biochemical relapse (defined as post-surgery PSA > 0.2 ng/ml; post-radiation > nadir +2 ng/ml, the PSA nadir is the lowest PSA reading achieved after treatment), with linear progression of at least 3 PSA tests in at least 3 months before the commencement of the trial.
* All patients must have negative bone scan and CT scan for the chest-abdomen-pelvis within 2 weeks prior to study initiation.

Exclusion Criteria:

* Psychological, familial, sociological or geographical conditions that may interfere with compliance with the study or prevent completion or compliance of protocol.
* Other severe or poorly controlled medical condition(s).
* Known allergies to any of the ingredients.
* Hormonal therapy or other therapy for PC in the last 3 months.
* Positive bone scan or CT scan of the chest-abdomen-pelvis.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-06; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Prostate Specific Antigen (PSA) kinetics in men with biochemical relapsed prostate cancer and serial increases in PSA levels. | 6 month endpoint.
  PSA doubling time increase will be used to show effectiveness of the Modified Citrus pectin (MCP).

SECONDARY OUTCOMES:
An assessment of adverse side effects due to Modified Citrus Pectin (MCP). | 6 month endpoint.
  Patient tolerability of MCP will be assessed by comparing the results of weekly self-assessment diaries with baseline assessments.

OTHER OUTCOMES:
Blood Serum Analysis (Galectin-3, C-Reactive Protein, Lipid Panels) | 6 month endpoint.
  At baseline (0 month), and end of study (6 month): Blood draw for serum levels of galectin-3, C-reactive protein, and lipid panel.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Keizman, MD, Principal Investigator — Genitourinary Oncology Service, Institute of Oncology, Meir Medical Center; Isaac Eliaz, MD, LAc, MS, Study Director — Amitabha Medical Clinic and Healing Center; Moshe Frenkel, MD, Study Chair — Clinical Associate Professor, University of Texas
Locations (1):
- Genitourinary Oncology Service, Institute of Oncology, Meir Medical Center, Tshernichovsky 59,, Kfar Saba, Israel

REFERENCES:
- [Background] Keizman D, Maimon N, Gottfried M. Metastatic hormone refractory prostate cancer: recent advances in standard treatment paradigm, and future directions. Am J Clin Oncol. 2014 Jun;37(3):289-96. doi: 10.1097/COC.0b013e318248dc1e. PMID 22772426
- [Background] Antonarakis ES, Zahurak ML, Lin J, Keizman D, Carducci MA, Eisenberger MA. Changes in PSA kinetics predict metastasis- free survival in men with PSA-recurrent prostate cancer treated with nonhormonal agents: combined analysis of 4 phase II trials. Cancer. 2012 Mar 15;118(6):1533-42. doi: 10.1002/cncr.26437. PMID 21960118
- [Background] Nangia-Makker P, Conklin J, Hogan V, Raz A. Carbohydrate-binding proteins in cancer, and their ligands as therapeutic agents. Trends Mol Med. 2002 Apr;8(4):187-92. doi: 10.1016/s1471-4914(02)02295-5. PMID 11927277
- [Background] Yan J, Katz A. PectaSol-C modified citrus pectin induces apoptosis and inhibition of proliferation in human and mouse androgen-dependent and- independent prostate cancer cells. Integr Cancer Ther. 2010 Jun;9(2):197-203. doi: 10.1177/1534735410369672. Epub 2010 May 11. PMID 20462856
- [Background] Kolatsi-Joannou M, Price KL, Winyard PJ, Long DA. Modified citrus pectin reduces galectin-3 expression and disease severity in experimental acute kidney injury. PLoS One. 2011 Apr 8;6(4):e18683. doi: 10.1371/journal.pone.0018683. PMID 21494626
- [Background] Ramachandran C, Wilk BJ, Hotchkiss A, Chau H, Eliaz I, Melnick SJ. Activation of human T-helper/inducer cell, T-cytotoxic cell, B-cell, and natural killer (NK)-cells and induction of natural killer cell activity against K562 chronic myeloid leukemia cells with modified citrus pectin. BMC Complement Altern Med. 2011 Aug 4;11:59. doi: 10.1186/1472-6882-11-59. PMID 21816083
- [Background] Jiang J, Eliaz I, Sliva D. Synergistic and additive effects of modified citrus pectin with two polybotanical compounds, in the suppression of invasive behavior of human breast and prostate cancer cells. Integr Cancer Ther. 2013 Mar;12(2):145-52. doi: 10.1177/1534735412442369. Epub 2012 Apr 24. PMID 22532035
- [Background] Liu HY, Huang ZL, Yang GH, Lu WQ, Yu NR. Inhibitory effect of modified citrus pectin on liver metastases in a mouse colon cancer model. World J Gastroenterol. 2008 Dec 28;14(48):7386-91. doi: 10.3748/wjg.14.7386. PMID 19109874
- [Background] Glinsky VV, Raz A. Modified citrus pectin anti-metastatic properties: one bullet, multiple targets. Carbohydr Res. 2009 Sep 28;344(14):1788-91. doi: 10.1016/j.carres.2008.08.038. Epub 2008 Sep 26. PMID 19061992
- [Background] Zhao ZY, Liang L, Fan X, Yu Z, Hotchkiss AT, Wilk BJ, Eliaz I. The role of modified citrus pectin as an effective chelator of lead in children hospitalized with toxic lead levels. Altern Ther Health Med. 2008 Jul-Aug;14(4):34-8. PMID 18616067
- [Background] Eliaz I, Weil E, Wilk B. Integrative medicine and the role of modified citrus pectin/alginates in heavy metal chelation and detoxification--five case reports. Forsch Komplementmed. 2007 Dec;14(6):358-64. doi: 10.1159/000109829. Epub 2007 Dec 12. PMID 18219211
- [Background] Johnson KD, Glinskii OV, Mossine VV, Turk JR, Mawhinney TP, Anthony DC, Henry CJ, Huxley VH, Glinsky GV, Pienta KJ, Raz A, Glinsky VV. Galectin-3 as a potential therapeutic target in tumors arising from malignant endothelia. Neoplasia. 2007 Aug;9(8):662-70. doi: 10.1593/neo.07433. PMID 17786185
- [Background] Eliaz I, Hotchkiss AT, Fishman ML, Rode D. The effect of modified citrus pectin on urinary excretion of toxic elements. Phytother Res. 2006 Oct;20(10):859-64. doi: 10.1002/ptr.1953. PMID 16835878
- [Background] Guess BW, Scholz MC, Strum SB, Lam RY, Johnson HJ, Jennrich RI. Modified citrus pectin (MCP) increases the prostate-specific antigen doubling time in men with prostate cancer: a phase II pilot study. Prostate Cancer Prostatic Dis. 2003;6(4):301-4. doi: 10.1038/sj.pcan.4500679. PMID 14663471
- [Background] Nangia-Makker P, Hogan V, Honjo Y, Baccarini S, Tait L, Bresalier R, Raz A. Inhibition of human cancer cell growth and metastasis in nude mice by oral intake of modified citrus pectin. J Natl Cancer Inst. 2002 Dec 18;94(24):1854-62. doi: 10.1093/jnci/94.24.1854. PMID 12488479
- [Background] Tehranian N, Sepehri H, Mehdipour P, Biramijamal F, Hossein-Nezhad A, Sarrafnejad A, Hajizadeh E. Combination effect of PectaSol and Doxorubicin on viability, cell cycle arrest and apoptosis in DU-145 and LNCaP prostate cancer cell lines. Cell Biol Int. 2012 Jul;36(7):601-10. doi: 10.1042/CBI20110309. PMID 22214228
- [Background] Hayashi A, Gillen AC, Lott JR. Effects of daily oral administration of quercetin chalcone and modified citrus pectin on implanted colon-25 tumor growth in Balb-c mice. Altern Med Rev. 2000 Dec;5(6):546-52. PMID 11134977
- [Background] Pienta KJ, Naik H, Akhtar A, Yamazaki K, Replogle TS, Lehr J, Donat TL, Tait L, Hogan V, Raz A. Inhibition of spontaneous metastasis in a rat prostate cancer model by oral administration of modified citrus pectin. J Natl Cancer Inst. 1995 Mar 1;87(5):348-53. doi: 10.1093/jnci/87.5.348. PMID 7853416
- [Background] Platt D, Raz A. Modulation of the lung colonization of B16-F1 melanoma cells by citrus pectin. J Natl Cancer Inst. 1992 Mar 18;84(6):438-42. doi: 10.1093/jnci/84.6.438. PMID 1538421
- [Background] Gunning AP, Bongaerts RJ, Morris VJ. Recognition of galactan components of pectin by galectin-3. FASEB J. 2009 Feb;23(2):415-24. doi: 10.1096/fj.08-106617. Epub 2008 Oct 2. PMID 18832596
- [Background] Azemar M, Hildenbrand B, Haering B, Heim ME, Unger C. Clinical benefit in patients with advanced solid tumors treated with modified citrus pectin: a prospective pilot study. Clin Med: Oncol. 2007;1:73-80.
- [Background] Calvier L, Miana M, Reboul P, Cachofeiro V, Martinez-Martinez E, de Boer RA, Poirier F, Lacolley P, Zannad F, Rossignol P, Lopez-Andres N. Galectin-3 mediates aldosterone-induced vascular fibrosis. Arterioscler Thromb Vasc Biol. 2013 Jan;33(1):67-75. doi: 10.1161/ATVBAHA.112.300569. Epub 2012 Nov 1. PMID 23117656
- [Background] Calvier L, Martinez-Martinez E, Miana M, Cachofeiro V, Rousseau E, Sadaba JR, Zannad F, Rossignol P, Lopez-Andres N. The impact of galectin-3 inhibition on aldosterone-induced cardiac and renal injuries. JACC Heart Fail. 2015 Jan;3(1):59-67. doi: 10.1016/j.jchf.2014.08.002. Epub 2014 Nov 11. PMID 25458174
- [Background] Dange MC, Srinivasan N, More SK, Bane SM, Upadhya A, Ingle AD, Gude RP, Mukhopadhyaya R, Kalraiya RD. Galectin-3 expressed on different lung compartments promotes organ specific metastasis by facilitating arrest, extravasation and organ colonization via high affinity ligands on melanoma cells. Clin Exp Metastasis. 2014 Aug;31(6):661-73. doi: 10.1007/s10585-014-9657-2. Epub 2014 Jun 21. PMID 24952269
- [Background] Hossein G, Keshavarz M, Ahmadi S, Naderi N. Synergistic effects of PectaSol-C modified citrus pectin an inhibitor of Galectin-3 and paclitaxel on apoptosis of human SKOV-3 ovarian cancer cells. Asian Pac J Cancer Prev. 2013;14(12):7561-8. doi: 10.7314/apjcp.2013.14.12.7561. PMID 24460334